CLINICAL TRIAL: NCT00665275
Title: The Use of Complementary and Alternative Medicine Among Outpatients With Inflammatory Rheumatic Diseases in Western Sweden.
Brief Title: Complementary and Alternative Medicine Among Outpatients With Inflammatory Rheumatic Diseases in Western Sweden
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Helena Forsblad d'Elia, Department of Rheumatology and Inflammation Research
Other Study IDs: VGFOUREG-8462; VGFOUREG-12277
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-04

CONDITIONS: Rheumatic Diseases
Keywords: complementary; alternative; medicine
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study aiming to study the use of complementary and alternative medicine (CAM) drugs and methods among patients with inflammatory rheumatic diseases, at Rheumatology clinics in western Sweden and also to investigate possible associations between CAM using habits and other characteristics of the patients.

DETAILED DESCRIPTION:
Complementary and alternative medicine (CAM) is treatment that primarily is given outside the institutions where conventional medicine is practised. CAM drugs are substances that often have a natural origin and are taken orally or used topically, for self-treatment. CAM methods are therapies where the patient often goes to a practitioner, for example acupuncture, massage, homeopathy or chiropractics.

Most cultures have their own history of traditional treatments, with herbal medicine or spiritual healers.

The use of complementary and alternative medicine (CAM) is widespread and increasing in many countries. The sales figures in Sweden for CAM drugs, functional foods and dietary supplements have increased from 450 million to 4250 million SEK between 1980 and 2007. Many people of today use CAM as a complement, rather than an alternative, to conventional healthcare. Some alternative methods, like acupuncture and massage, have also been integrated into conventional medicine.

The biological effects of drugs containing herbs or animal parts are often unknown and there is a hazard of interaction with prescribed medication.

The use of CAM drugs is often not communicated by the patient to the physician. A Swedish point observation study of patients admitted to Sahlgrenska hospital 2004 showed that 69 % of the patients had used CAM drugs at any time in their life, but only 27,5% had informed their doctor about it. The use of CAM drugs was seldom documented in the medical records of the patient.

The utilization of CAM among patients with rheumatic diseases in Sweden has never been studied before.

The aim of this trial was to study the use of CAM methods and CAM drugs among patients seen at rheumatology practises in the west of Sweden. To investigate which methods and drugs that are being used and to see if there are connections between using habits and factors like gender, age, rheumatic diagnoses, disease activity, medication and the patients experience of pain, fatigue and general health. We were also interested in finding out the reason for use of CAM, and if the patients had experienced beneficial effects or side effects of the use.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for inclusion if they were attending the rheumatology clinic and had had an appointment there before.

Exclusion Criteria:

* Patients were excluded if they were on their first visit to the practice, had dementia or had difficulties understanding Swedish.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lists of outpatients who were scheduled for appointments at the rheumatology clinic were sent to an external randomizer, to randomly elect patients who were asked to participate. Patients were eligible for inclusion if they were attending the rheumatology clinic and had had an appointment there before. Patients were excluded if they were on their first visit to the practice, had dementia or had difficulties understanding Swedish.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The prevalence of complementary and alternative medicine (CAM) drugs and methods among patients with inflammatory rheumatic diseases in western Sweden. | July 2007

SECONDARY OUTCOMES:
To investigate potential significant associations between CAM using habits and characteristics of the patients. | July 2007

CONTACTS AND LOCATIONS:
Overall Officials: Helena Forsblad d'Elia, MD, PhD, Principal Investigator — Department of Rheumatology and Inflammation Research, Sahlgrenska Academy at University of Gothenburg
Locations (1):
- Department of Rheumatology, Sahlgrenska University Hospital, Gothenburg, Sweden